CLINICAL TRIAL: NCT04860843
Title: Regional Nerve Blocks in Alloplastic Breast Reconstructive Surgery: A Pilot, Randomized Controlled Trial
Brief Title: Nerve Blocks in Alloplastic Breast Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kathryn Isaac, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H20-00787
Record Dates: First submitted 2020-12-16; First posted 2021-04-27 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Surgery, Plastic; Mastectomy; Nerve Block; Breast Reconstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local anesthetic TPVB + Local anesthetic Pecs block (Experimental): Patients will receive a thoracic paravertebral with pecs block, both with local anesthetic infiltrate.
  Interventions: Drug: Thoracic paravertebral block; Drug: Pecs block
- Local anesthetic TPVB + Sham Pecs block (Sham Comparator): Patients will receive a thoracic paravertebral with local anesthetic infiltrate and a pecs block with saline infiltrate.
  Interventions: Drug: Thoracic paravertebral block; Drug: Sham Pecs block

INTERVENTIONS:
Drug: Thoracic paravertebral block — Participants will receive a thoracic paravertebral with local anesthetic infiltrate (30ml of 0.35% ropivacaine with 1:400K epinephrine).
Drug: Pecs block — Participants will receive a pecs block with local anesthetic infiltrate (30ml of 0.25% ropivacaine with 1:400K epinephrine).
  Arms: Local anesthetic TPVB + Local anesthetic Pecs block
Drug: Sham Pecs block — Participants will receive a and a pecs block with saline infiltrate (30ml normal saline; 0.9% NaCl).
  Arms: Local anesthetic TPVB + Sham Pecs block

SUMMARY:
Pain management is a major concern in oncologic breast surgery and reconstruction. Significant risks for acute and chronic pain after surgery might be reduced through improved pain control pre-operatively. Addition of regional anesthesia to a multimodal peri-operative pain management protocol offers a promising solution for improved recovery. For patients undergoing mastectomy with immediate alloplastic breast reconstruction, this RCT compares TPVB+Pecs local anesthetic block with TPVB local anesthetic block and Pecs placebo normal saline block for their effect on acute pain, chronic pain, opioid consumption, opioid-related side effects, patient-reported quality of recovery after surgery, and length of stay.

DETAILED DESCRIPTION:
OBJECTIVES

The primary objectives of the pilot trial are to demonstrate feasibility of recruitment and to demonstrate efficacy potential. The primary objectives of the definitive trial are to determine if Thoracic Paravertebral with Pecs blocks (defined as Pec I and Pec II blocks) (TPVB+Pecs) will reduce opioid consumption and chronic pain compared to a TPVB+Sham block in patients undergoing mastectomy with IBR using tissue expanders or implants. Secondary objectives of the definitive trial include assessment of opioid consumption, patient-reported postoperative pain scores, postoperative nausea and vomiting, length of stay, and patient-reported quality of recovery.

HYPOTHESIS

In breast cancer patients undergoing mastectomy with immediate implant-based breast reconstruction, the addition of a Pecs block to a thoracic paravertebral block (TPVB+Pecs) will reduce acute and chronic patient-reported postoperative pain as compared to a thoracic paravertebral block with sham Pecs block (TPVB+Sham).

Secondary hypotheses include: the TPVB+Pecs over TPVB+Sham will decrease opioid consumption, postoperative nausea and vomiting, decrease patient-reported postoperative pain scores, length of stay, and improve patient-reported quality of recovery in patients undergoing total mastectomy with IBR using tissue expanders or immediate implants.

JUSTIFICATION

The definitive trial will determine if TPVB+Pecs improves postoperative acute and chronic pain and reduces opioid use for patients undergoing mastectomy with IBR using tissue expanders or immediate implants.

International Consensus guidelines for ERAS in breast reconstruction make a strong recommendation for multimodal, opioid-sparing analgesia postoperatively based on high-level evidence. Increased total opioid analgesic use has been shown to increase length of stay in hospital. Reduced opioid consumption results in less postoperative nausea, vomiting, and constipation, supports early ambulation, shortens hospital stays, and improves psychological well being. Current ERAS protocols for alloplastic breast reconstruction are successfully opioid-sparing and address acute recovery. However, opioids continue to play an important role in peri-operative protocols for achieving adequate pain control, which suggests further adjunctive strategies may be beneficial. Furthermore, the effects of peri-operative protocols on the development of chronic pain are lacking. By evaluating the effectiveness of TPVB+Pecs in alloplastic reconstruction, our proposed study would help to establish an important additional feature to the ERAS pathway for our hospital and other institutions.

STUDY DESIGN

The design of the pilot RCT is the same as the future definitive trial, a parallel-group, double-blinded RCT. The target population includes patients undergoing mastectomy with IBR using tissue expanders or immediate implants.

The study will compare two arms:

1. TPVB using local anesthetic infiltrate with Pecs using local anesthetic infiltrate (TPVB+Pecs, the intervention arm).

   OR
2. TPVB using local anesthetic infiltrate with Pecs using normal saline infiltrate (TPVB+Sham, the control arm).

The pilot trial will be conducted at Mount Saint Joseph Hospital (MSJH). The assignment of intervention will be determined by randomization through REDCap.

Each participant will be assigned a consecutive Study ID at time of enrollment. Patients will be randomized 1:1 to either TPVB+Pecs or TPVB+Sham. Patients undergoing symmetrizing procedures as part of a bilateral breast surgery will not have a regional block on the symmetrizing side (which is not IBR). Patients undergoing bilateral IBR surgery using implants or expanders on both breasts will not be included in the study due to risk of local anesthetic toxicity with bilateral TPVB.

The randomization sequence will be created using REDCap-generated 1:1 randomization with permuted blocks of varying size (4 and 6). The assignments (TPVB+Pecs or TPVB+Sham) will be placed in order in opaque, consecutively numbered envelopes. The sequence and envelopes will be created by an independent research assistant who will not be involved in the remainder of the study implementation.

Study participants, Operating Room (OR) anesthesiologists, surgeons, research assistants, and nurses in the OR, Post-anesthesia Care Unit (PACU), and ward will be blinded as to whether a participant receives TPVB+Pecs or TPVB+Sham block. At MSJH, the anesthesiologists in the operative theater are separate from the team of regional anesthesiologists performing regional blocks in the preoperative area. Only the regional anesthesiologist and anesthesia assistant in the preoperative block area, who will administer the regional block, will be unblinded.

On the day of surgery, the regional anesthesiologist at MSJH will be provided with the Study ID specific sealed envelope which will assign the patient to receive either the TPVB+Pecs or TPVB+Sham block. The regional anesthesiologist will prepare local anesthetic or normal saline injections for infiltration based on the random assignment. For all patients, the regional block will be performed as outlined in the Procedure Protocols (See Appendix 1: Nerve Block). All participants will receive general anesthesia following the nerve block. All other parameters and protocols will be identical.

Currently, at MSJH, approximately 4 - 5 cases of mastectomy with IBR are performed per week. We do not anticipate difficulty with enrolment into this study. This internal pilot will generate initial recruitment data to enable an early review and validation of our recruitment projections and study population target prior to transition to formal RCT.

Additional Details of Study Design

Participants will also be given at the time of consent a post operative package. This will contain the Quality of Recovery-15 Questionnaire (Form 7), Recovery Booklet (Form 5) and Pain Burden Index (Form 8).

The Quality of Recovery-15 Questionnaire (see Form 7) is to be completed at 24 hours after surgery in paper format or electronic format (based on their preference). This 24 hour time point will be marked on the QoR-15 form. If paper format is preferred, the QoR-15 will be provided with a paid-postage envelope to return once completed at 24 hours after surgery. The pain NRS at 24 hours will be recorded from the chart. The envelopes will be addressed to the research coordinator at UBC Hospital office. If the participant prefers electronic format, the questionnaire will be sent to their provided email address using secure online format (REDCap developed questionnaire).

Recovery Booklet (see Form 5) will include: a) schedule for taking prescription pain medications; b) a postoperative 7-day symptom diary (for recording pain on NRS at 24 hours, episodes of vomiting, nausea, and use of prescribed medications). Patients will be provided with a paid-postage envelope to return their Recovery Booklet via mail once completed 7 days after surgery. Patients will be reminded to complete the Recovery Booklet (Form 5) in 3-4 days and once again at 14 days to return the envelope.

The Pain Burden Index questionnaire (see Form 8) asks specifically about pain in four surgically related body areas and to calculate the Pain Burden Index (PBI). The PBI is calculated by summing the pain severity scale (0-10) at each of four locations (breast, axilla, chest wall, arm) multiplied by the frequency of the pain at each site. The PBI questionnaire will be sent to participants via mail as paper format (with paid-postage envelope to return once completed) or email as electronic format (as per their requested preference) to be completed 3 and 6 months after their surgery. Details of present adjuvant treatments (radiation and chemotherapy) will also be included in the questionnaire.

Secondary outcomes data including opioid consumption and side effects, length of stay in hospital (hours), rescue medications, failure of early discharge, complications and adverse events and time-based outcome measures (time in PACU, time under general anesthesia, time to perform ultrasound-guided TPVB+PecsII, failure of discharge from PACU and requiring admission) will be collected through participants' charts and EMR.

STATISTICAL ANALYSIS

Patient characteristics and outcome measures will be summarized by group. An 80% confidence interval for the difference in average pain score over 24 hours will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be female, and at least 19 years old.
2. Patients must be ASA grade I or II.
3. Patients must be undergoing total mastectomy with IBR using tissue expander or implant, with or without axillary surgery.

Exclusion Criteria:

1. Patients have a known contraindication for a regional block: known coagulation disorder, treatment with anticoagulants, infection at the injection site, known allergy to medication in the study.
2. Patients who are pregnant at the time of surgery.
3. Patients having bilateral mastectomy and immediate alloplastic breast reconstruction (as only one side can be blocked to prevent local anesthesia toxicity).
4. Patients with ASA Class III or IV.
5. Patients with BMI>35kg/m2.
6. Patients weighing less than 50kg.
7. Patients living/staying outside of 1-hour driving distance from hospital.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Rate of participant recruitment | 1 year
  The definitive trial will be considered feasible if > 50% of eligible patients are enrolled in this pilot study.
Rate of successful nerve blocks | 1 year
  The definitive trial will be considered feasible if > 90% of blocks are successful.
Rate of participant retention | 6 months
  The definitive trial will be considered feasible if there is > 90% participant retention at 6 months.
Average pain score in the 24-hour post-operative period assessed by the Numerical Rating Scale. | 24 hours post-operatively
  The Numerical Rating Scale is an 11-point scale (0-10), where a lower number indicates less pain. We will consider preliminary evidence of efficacy for a definitive trial if the 80% confidence interval for the between-group difference in average pain score in the 24-hour postoperative period favours LA block.

SECONDARY OUTCOMES:
Opioid analgesia requirements | 24 hours post-operatively
  Will include intraoperative opioids administered in the OR and postoperative opioids administered/ingested in the Postanesthetic Care Unit (PACU), Surgical Day Care Unit (SDC), Inpatient Unit, and home in the 24-hour period after completion of surgery. Opioids consumed will be converted to MME.
Acute patient-reported pain scores assessed by the Numerical Rating Scale | Up to 24 hours post-operatively
  The Numerical Rating Scale is an 11-point scale (0-10), where a lower number indicates less pain). It will be measured at the standard time points of nursing care assessments: preoperatively (baseline); four times per hour in PACU until discharge; if admitted, hourly for 2 hours, and then every 6 hours in the Inpatient Unit; and at discharge from hospital; 24 hours after surgery is complete.
Post-operative nausea measured by the Numerical Rating Scale | 24 hours post-operatively
  The Numerical Rating Scale is an 11-point scale (0-10), where a higher score indicates a better outcome/ less nausea.
Post-operative vomiting measured by number of vomiting episodes | Up to 48 hours post-operatively
  Number of vomiting episodes in the post-anesthesia care unit and at home will be measured.
Quality of Recovery Score measured by the Quality of Recovery 15 Questionnaire | Baseline (prior to surgery) and 24 hours after surgery
  The Quality of Recovery 15 (QoR-15) is a 15-item questionnaire that assesses patient-reported pain, physical comfort, physical independence, psychological support, and emotional state. Questions are rated in an 11-point scale (0-10), where a higher score indicates a better outcome. The QoR-15 takes an average of 2.5 minutes to complete. The QoR-15 has been statistically validated and is designed for both ambulatory and inpatient surgery populations. The QoR-15 will be completed at baseline prior to surgery and 24 hours after surgery.
Length of stay in hospital in hours | Up to 96 hours post-operatively
  Measured from the time admitted to PACU to the time discharged from hospital. LOS includes time in the PACU, Surgical Day Care (SDC) and, if required, Inpatient Unit. Patients are transferred between units and discharged from hospital according to standardized institutional criteria
Time to perform ultrasound-guided TPVB+PecsII | Up to 24 hours post-operatively
  Measured in minutes.
Time under general anesthesia | Up to 24 hours post-operatively
  Measured in minutes.
Time in PACU | Up to 24 hours post-operatively
  Measured in minutes.
Number of participants with failure of discharge from PACU and requiring admission to hospital | Up to 24 hours post-operatively
  Categorical.
Number of participants requiring rescue opioid analgesics and anti-emetics. | Up to 7 days post-operatively
  Rescue medication are defined as those required "as needed" (ie. Beyond scheduled) in the PACU, ward and after discharge.
Time to rescue opioid analgesics and anti-emetics. | Up to 7 days post-operatively
  Rescue medication are defined as those required "as needed" (ie. Beyond scheduled) in the PACU, ward and after discharge. Time to rescue medications is measured in minutes.
Number of participants with failure of early discharge. | Up to 48 hours post-operatively
  Failure of early discharge is defined as emergency room visits within 48 hours of discharge
Number of participants with complications and adverse events | Up to 24 hours post-operatively
  Related to the ultrasound-guided regional block: vascular or nerve injury, Horner's syndrome, bleeding/hematoma, local anesthetic systemic toxicity, pneumothorax, distortion tissue planes during axillary dissection, and other.
  Related to the surgery: hematoma, tissue necrosis, urgent unplanned return to the operative theater within 24 hours of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Isaac, MD MPH FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- Mount St Joseph Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Wells H, Malik K, Brasher PMA, Bovill E, Van Laeken N, Warburton R, Prabhakar C, Li XL, Isaac KV. The addition of interpectoral and pectoserratus fascial plane blocks to paravertebral blocks for analgesia after total mastectomy and immediate breast reconstruction: a pilot feasibility randomized controlled trial. Can J Anaesth. 2025 Sep;72(9):1387-1396. doi: 10.1007/s12630-025-03030-1. Epub 2025 Sep 22. PMID 40983823

DOCUMENTS (1):
  • Study Protocol (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT04860843/Prot_000.pdf